CLINICAL TRIAL: NCT05492890
Title: The Use of Continuous Glucose Monitors in the Intrapartum and Postpartum Inpatient Care of Women With Diabetes Mellitus: A Randomized Noninferiority
Brief Title: Continuous Glucose Monitoring for Women With Diabetes Mellitus in the Intrapartum and Postpartum Inpatient Care
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020H0498
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Diabetes, Gestational
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Point of care blood glucose samples will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Dexcom CGM: Continuous glucose monitoring
  Interventions: Device: Dexcom G6
- Point of care testing: Finger poke glucose measure

INTERVENTIONS:
Device: Dexcom G6 — Continuous glucose monitoring
  Groups: Dexcom CGM

SUMMARY:
Diabetes mellitus affects roughly 8% of pregnancies and is associated with significant perinatal and maternal morbidity. Increasing numbers of women are either entering pregnancy with a continuous glucose monitor (CGM) or are initiating use during pregnancy, with data emerging suggesting improved outcomes among those using CGM. Since the introduction of CGM in the late 1990s, there has been slow acceptance of their validation and use in the inpatient setting. The investigators propose an observational prospective cohort study to analyze the correlation of CGM data with traditional capillary glucose readings in the intrapartum and postpartum settings.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* Women with a viable singleton or twin intrauterine pregnancy between 22 5/7 and 41 6/7 weeks gestation based on the best obstetric estimate by ACOG criteria
* Diagnosis of insulin-dependent pregestational diabetes mellitus (type 1 or type 2 diabetes)
* Planning to deliver at OSU Wexner Medical Center
* Able to understand the study, and having understood, provide written informed consent in English

Exclusion Criteria:

* Gestational diabetes mellitus, Maturity Onset Diabetes of Young, and Cystic Fibrosis Related Diabetes
* Abnormal obstetrical ultrasound suspicious for major congenital abnormality
* Known or suspected fetal aneuploidy (by either CVS, amniocentesis, or cell-free DNA)
* Participation in another trial that may influence the primary outcome, without prior approval
* Participation in this trial in a prior pregnancy
* Higher order pregnancy
* History of severe skin allergy to adhesive products or CGM within the previous 3 months

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Pregnant woman
Study Population: Women ages 18-45 who are pregnant
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Maternal outcome | 9 months
  Assessed by analyzing the number of hypoglycemic and hyperglycemic episodes prior to and post-delivery as determined by glucose measurements

SECONDARY OUTCOMES:
Neonatal outcomes | 10 days
  Assessed by requirement of neonatal antidiabetic care measured in the number of hypoglycemic episode requiring IV dextrose treatment

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Buschur, MD, Principal Investigator — tOSU Medical Center

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with outside investigators